CLINICAL TRIAL: NCT04553887
Title: Almonertinib as Upfront Treatment for Uncommon EGFR Mutation Harboring Non-Small-Cell Lung Cancer Patients: A Multicenter, Open-Label, Phase II Trial
Acronym: AUTUMN
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTUMN
Record Dates: First submitted 2020-09-12; First posted 2020-09-18 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Previously treated NSCLC patients with EGFR exon 20 insertion mutantion
  Interventions: Drug: Almonertinib
- Cohort 2 (Experimental): NSCLC Patients with uncommon EGFR Mutation
  Interventions: Drug: Almonertinib

INTERVENTIONS:
Drug: Almonertinib — single agent, 110mg p.o once daily until disease progressed

SUMMARY:
This is a Phase 2 study to evaluate the efficacy and the safety/ tolerability of Almonertinib in NSCLC patients with uncommon EGFR Mutation or EGFR exon 20 insertion mutations. Patients with EGFR exon 20 insertion mutations have to had at least one prior systemic treatment for locally advanced or metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75years#ECOG PS#0-2#Life expectancy of more than 3 months#with measurable lesion ( RECIST1.1).
2. Cohort A: Patients with EGFR exon 20 insertion, failure of first-line standard chemotherapy, or intolerance to chemotherapy Cohort B: Patients with uncommen EGFR mutations but without exon 19 deletion, L858R, T790M, and exon 20 insertion
3. ≥1 target lesion that has not received radiotherapy in the past 3 months and can be accurately measured in at least 1 direction#Previously received radiation therapy, but the radiotherapy area must be <25% of the bone marrow area, and radiation therapy must have closed for at least≥4 weeks at the time of enrollment.
4. Main organs function is normal.
5. Signed and dated informed consent.

Exclusion Criteria:

1. Patient has had previous treatment with Pyrotinib, Poziotinib or any other EGFR or HER2 exon 20 insertion mutation-selective tyrosine kinase inhibitor (TKI) prior to study participation. The currently approved TKIs (ie, erlotinib, gefitinib, afatinib, osimertinib) are not considered to be exon 20 insertion-selective and are permissible

1. Patients with EGFR 19 exon deletion mutation, 21 exon L858R mutation or 20 exon T790M mutation.
2. Small cell lung cancer (including mixed small cell and non-small cell lung cancer);
3. Cohort A: Patients who had previously used the third generation of EGFR-TKI (including Almonertinib, Osimertinib, etc.) Cohort B: Patients who had previously used EGFR-TKI
4. Patients who planned to receive systemic anti-tumor therapy within 4 weeks prior to allocation or during the course of this study, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or receiving the Mitomycin C 6 weeks prior to medication). Extra-field radiotherapy (EF-RT) was performed 4 weeks prior to allocation or restricted radiotherapy for assessing tumor lesions within 2 weeks prior to allocation
5. With kinds of factors which affect oral medicine (e.g. failing to swallow, gastrointestinal tract getting resected, chronic diarrhea and ileus)
6. Subjects with uncontrolled hypokalemia and hypomagnesemia before study entry
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Almonertinib
8. History of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease, or history of organ transplantation; active infection including hepatitis B (HBV DNA level ≥1000 copies /mL), hepatitis C and human immunodeficiency virus (HIV); Severe acute or chronic infections requiring systemic treatment
9. Subjects had any heart disease, including: (1) angina; (2) requiring medication or clinically significant arrhythmia; (3) myocardial infarction; (4) heart failure; (5) Any heart diseases judged by investigator as unsuitable to participate in the trial
10. Known history of neurological or psychiatric disease, including epilepsy or dementia
11. Has a history of malignant tumors. Except for patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or orthotopic cervical cancer who have undergone curative treatment and have no disease recurrence within 5 years after the start of treatment
12. Respiratory syndrome (dyspnea≥CTC AE 2), severe pleural effusion, ascites, pericardial effusion
13. Patient has had other malignancies within the past 3 years, except for stable non-melanoma skin cancer, fully treated and stable early stage prostate cancer or carcinoma in situ of the cervix or breast without need of treatment
14. Patient is pregnant or breast-feeding
15. Judgment by the investigator that should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | To evaluate objective response rate 6-8 weeks after the initiation of Almonertinib
  The proportion of subjects who achieve Complete Response (CR) and Partial Response (PR) by the best response from the first dose of Almonertinib to the end of study.

SECONDARY OUTCOMES:
Progression Free Survival | 30 months
  The PFS time is defined as time from enrollment to locoregional or systemic recurrence, second malignancy or death due to any cause; censored observations will be the last date of : "death", "last tumor assessment", "last follow up date" or "last date in drug log"
Disease Control Rate | 30 months
  Disease Control Rate (DCR) defined as the percentage of participants with Disease Control best overall response (complete response, partial response or stable disease).
Overall Survival | 30 months
  OS was defined as time from date of enrollment to date of death due to any cause. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.
Duration of Response | 30 months
  Number of days from the date that measurement criteria are first met for CR or PR (whichever status is recorded first) until the first subsequent date that progressive disease or death is documented.
Safety and Tolerability | 30 months
  Number of Participants with treatment related Adverse Events as Assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Dingzhi Huang, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Identified individul participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external indepentent Review Panel. Requestors will be required to sign a Data Access Agreement.